CLINICAL TRIAL: NCT03387787
Title: Pilot Study to Evaluate Glycaemic Control Using GlucoTab® With Insulin Degludec and Aspart in Hospitalized Patients With Diabetes Mellitus Type 2
Brief Title: Evaluation of Glycaemic Control Using GlucoTab® With Insulin Degludec in Hospitalized Patients With Diabetes Mellitus Type 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDEM_GlucoTab
Record Dates: First submitted 2017-12-15; First posted 2018-01-02 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: GlucoTab, Tresiba, Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GlucoTab Treatment Arm (Experimental): Recruited patients will be treated with insulin degludec and insulin aspart. insulin doses will be calculated by the GlucoTab system
  Interventions: Device: GlucoTab; Drug: Insulin Degludec

INTERVENTIONS:
Device: GlucoTab — The GlucoTab® system is a computerized decision support system built of an android based front-end user interface and a backend server including the REACTION algorithm. GlucoTab® is able to process blood glucose data and physiological confounders of glycaemia. Subsequently, GlucoTab® provides patient-specific basal, bolus, and correction insulin doses together with visualization and documentation of relevant data.
  Insulin doses of recruited patients will be calculated by the GlucoTab System for at least 48 hours and a maximum duration of 21 days.
Drug: Insulin Degludec — During the study, patients will be treated with basal Insulin degludec

SUMMARY:
The GlucoTab® system is a computerized decision support system built of an android based front-end user interface and a backend server including the REACTION algorithm. GlucoTab® is able to process blood glucose data and physiological confounders of glycaemia. Subsequently, GlucoTab® provides patient-specific basal, bolus, and correction insulin doses together with visualization and documentation of relevant data. The GlucoTab® system was found capable to keep hospitalized diabetic patients in the recommended target range without increasing the risk for hypoglycaemic events. Insulin pharmacokinetic is a critical confounder of glycaemic variability and the main determinant of an algorithm-based decision support-system. GlucoTab® is intended for being used with a basal/bolus insulin regimen. Up to date, feasibility data are limited to the use of insulin glargine.

Insulin degludec, an ultra-long acting basal insulin is characterized by a stable pharmacokinetic profile a half-life of ~25 hours. It was found equally effective to insulin glargine with respect to glycaemic control, while the incidence of (nocturnal) hypoglycaemia was smaller in patients treated with insulin degludec. Within the present study, insulin glargine will be replaced by insulin degludec, which is not yet approved for dose titration with GlucoTab®.

In the present study, 15 non-critically ill T2DM patients, who were hospitalized at the University Clinic of Neurosurgery for various reasons and require insulin treatment will be recruited. Patients will be treated with insulin Tresiba and insulin Novorapid. For a maximum duration of 21 days, GlucoTab® will calculate the required insulin doses for each patient, depending on fasting plasma glucose and postprandial glucose measurements during the day. After the calculated Insulin dose has been approved by the physician, the nursing staff will give the dose to the respective patient.

The present study will analyse the efficacy of GlucoTab® for glycaemic management in T2DM patients using insulin degludec.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent after being advised of every detail of the study
* Male or female sex
* Aged ≥ 18 years
* Known history of diabetes of at least 90 days
* Type 2 diabetes mellitus treated with either diet alone or any combination of oral antidiabetic agents and the absence of diabetic ketoacidosis for at least 90 days.
* HbA1c 6.5 - 10.0%

Exclusion Criteria:

* Type 1 diabetes mellitus
* Gestational diabetes mellitus
* Pregnancy or currently breast-feeding women
* Known or suspected allergy to insulin degludec and/or insulin aspart
* Continuous parenteral nutrition
* Participation in another trial which may in the opinion of the investigator interfere with the software algorithm
* Any mental condition rendering the patient incapable of giving informed consent
* Any disease or condition which in the opinion of the investigator would interfere with the trial performance and/or the physical and/or psychosocial safety of the study participant
* Critically ill patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Blood Glucose in target range in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
  We measure mean percentage of blood glucose measurements in the target range of ≥5.6 mmol/l ≤7.8 mmol/l.
Random blood glucose <9.9 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
  We measure random daily blood glucose concentrations <9.9 mmol/l as calculated by all pre-prandial and bedtime glucose values measured ≥24 hours after start of insulin therapy

SECONDARY OUTCOMES:
Number of severe hypoglycaemic episodes (defined as symptomatic or asymptomatic hypoglycaemia requiring third party help) | during the treatment period (at least 48 hours but maximal 21 days per patient)
Number of overall hypoglycaemic episodes defined as any measurement of capillary glucose concentrations ≤3.9 mmol/l with or without symptoms related to low blood glucose, according to the current definition of the American Diabetes Association (ADA) | during the treatment period (at least 48 hours but maximal 21 days per patient)
Number of blood glucose measurements per day | during the treatment period (at least 48 hours but maximal 21 days per patient)
Number of missed blood glucose measurements | during the treatment period (at least 48 hours but maximal 21 days per patient)
Number of additionally required blood glucose measurements | during the treatment period (at least 48 hours but maximal 21 days per patient)
Correction factor insulin dose per day | during the treatment period (at least 48 hours but maximal 21 days per patient)
  As calculated by GlucoTab
Basal factor insulin dose per day | during the treatment period (at least 48 hours but maximal 21 days per patient)
  As calculated by GlucoTab
Bolus insulin dose per day | during the treatment period (at least 48 hours but maximal 21 days per patient)
  As calculated by GlucoTab
Number of insulin injections per day | during the treatment period (at least 48 hours but maximal 21 days per patient)
Number and reasons for non-performance of insulin injections per day | during the treatment period (at least 48 hours but maximal 21 days per patient)
Adherence to the insulin dose suggestion of the GlucoTab® system | during the treatment period (at least 48 hours but maximal 21 days per patient)
Mean daily blood glucose as calculated by pre-meal and bedtime blood glucose values: Overall and per treatment day | during the treatment period (at least 48 hours but maximal 21 days per patient)
Mean pre-bedtime blood glucose | during the treatment period (at least 48 hours but maximal 21 days per patient)
Mean pre-breakfast blood glucose | during the treatment period (at least 48 hours but maximal 21 days per patient)
Mean pre-lunch blood glucose | during the treatment period (at least 48 hours but maximal 21 days per patient)
Mean pre-dinner blood glucose | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose <2.2 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose between 2.201-<3.9 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose between 3.901-<5.5 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose between 5.501- <7.8 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose between 7.801-< 9.9 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose between 9.901-<16.6 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Blood glucose ≥16.601 mmol/l in percent | during the treatment period (at least 48 hours but maximal 21 days per patient)
Time of glucose measurements derived from CGM in the following ranges: 0-<2.2 mmol/l, 2.201-<3.9 mmol/l, 3.901-<5.5 mmol/l, 5.501-<7.8 mmol/l, 7.801-<9.9 mmol/l, 9.901-<16.6 mmol/l, ≥16.601 mmol/l | during the treatment period (at least 48 hours but maximal 21 days per patient)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Laimer, Prof. MD, Principal Investigator — Division of Endocrinology, Diabetes, Clinical Nutrition & Metabolism, Universitsy Hospital Bern, Switzerland
Locations (1):
- Division of Endocrinology, Diabetes, Clinical Nutrition & Metabolism, University Hospital Berne, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University Clinics of Neurosurgery — https://neurochirurgie.insel.ch/
- See also: The developers Homepage — http://www.glucotab.at/de/